CLINICAL TRIAL: NCT05922462
Title: Effects of Increased Greek Yogurt Consumption on Circulating Markers of Bone Metabolism and Inflammation in Youth and Young Adult Athletes
Brief Title: Effects of Increased Greek Yogurt Consumption in Youth and Young Adult Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: York University (Other)
Responsible Party: Principal Investigator, Panagiota Klentrou, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB 22-303
Record Dates: First submitted 2023-06-04; First posted 2023-06-28 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Bone Growth Abnormal; Inflammation
Keywords: Athletes; Bone markers; Inflammatory cytokines; Greek yogurt; Whey protein
MeSH Terms: conditions — Bone Diseases, Developmental; Inflammation | interventions — Whey Proteins

STUDY DESIGN:
Intervention Model Description: The study will use a randomized controlled parallel design, where participants will be randomly assigned to either to consume greek yogurt or whey protein for 16 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Greek yogurt intervention group (GY) (Experimental): Participants in the GY group will be instructed by a registered dietician to consume 2 servings/day (preferably morning and night) of 175 g GY (0% MF, flavoured, 130 calories, 17 g protein, 225 g calcium; e.g., OIKOS High Protein GY) for a total of 16 weeks. For their convenience, the athletes will be provided with appropriate scoops to measure out 175 g of GY per serving of the larger 650 g commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the feasibility of the intervention, the timing of the servings will be flexible to facilitate the training and competition routines. For the same reasons, the athletes will be able to choose the flavour of their GY.
  Interventions: Dietary Supplement: Greek yogurt
- Whey protein intervention group (WP) (Experimental): Participants in the WP group will follow a similar consumption schedule but will be instructed by the RD to consume two servings/day (preferably morning and night) each of 2/3 of a scoop of commercially available WP powder (flavoured, ~29 g, 120 calories, 19 g protein, 112.5 g calcium; e.g., PURE Whey Protein, Walmart) for a total of 16 weeks. The WP scoop will be dissolved in water (e.g., 1 g of WP isolate to 10 mL of water, as recommended by the manufacturer). This protein dose is similar to the previous dose in young swimmers and comparable to other studies in adults. Athletes will be provided with appropriately marked scoops (corresponding to 2/3 of the manufacturer scoop) to measure their single servings. Each athlete will receive two large containers (2 x 907 g = 1814 g per week) at the beginning of each week, which will be enough to cover the two daily servings of 29 g (i.e., 58 g/day).
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Greek yogurt — For 16 weeks, athletes will consume 2 servings/day of 175 g GY (0% MF, flavoured, 130 calories, 17 g protein, 225 g calcium; e.g., OIKOS High Protein GY)
  Arms: Greek yogurt intervention group (GY)
Dietary Supplement: Whey protein — For 16 weeks, athletes will consume 2 servings/day of 2/3 of a scoop of commercially available WP powder (flavoured, ~29 g, 120 calories, 19 g protein, 112.5 g calcium; e.g., PURE Whey Protein, Walmart)
  Arms: Whey protein intervention group (WP)

SUMMARY:
Physical activity and dairy consumption during growth and development are each known to improve peak bone mass in young adults. Peak bone mass, the maximum amount of bone a person will have in their lifetime, is typically reached in the early 20's in females and late 20's in males. However, evidence suggests that young people do not consume enough dairy to maximize their bone mass. The resulting effect in peak bone mass can be troublesome, particularly for athletes, such as volleyball players. This study aims to determine whether increased dairy consumption combined with training can have an additive effect on the physiology of young competitive athletes. Specifically, we will examine whether Greek yogurt consumption will lead to beneficial changes in bone metabolism and inflammation, in adolescent and young adult, male and female athletes, similar to those observed with whey protein supplementation. Many athletes choose exclusively protein supplementation and miss out on other nutrients vital for healthy growth and development. By examining the benefits of Greek yogurt across different athlete age groups and sexes, this work will help reshape the attitudes, beliefs, and behaviours surrounding diet of young athletes.

DETAILED DESCRIPTION:
Purpose: This study will investigate the effect of chronic high-impact exercise training and GY consumption on bone metabolism and inflammation compared with isonitrogenous/isocaloric whey protein (WP) supplementation (a common practice by athletes) in youth and young adult athletes.

Participants: A total of 40 varsity athletes (aged 17-22 years; 20 males, 20 females) will be recruited in year one, and 40 club athletes (aged 15-16 years; 20 males, 20 females) will be recruited in year two. Participants will be recruited from the varsity teams at Brock and club teams in the Niagara area (one male and one female team from each age group). All participants (and the parents/guardians of club athletes) will provide written informed consent in order to be included in the study. Potential participants will complete an online health screening questionnaire to document general health and individual and family health history. It will also be used to record information on medication use and for female participants to report menstrual history and status, as well as the use and type of oral contraceptives (brand and hormone). Athletes will be excluded from the study if they are injured and unable to participate in practices, have an allergy to dairy foods/dairy protein or have been diagnosed with lactose intolerance.

Athletes from each team will be randomly assigned to either the GY intervention group or the WP comparison group. Thus, eight treatment groups (n = 10 athletes per group):

* GY x Female Varsity
* GY x Male Varsity
* GY x Female Club
* GY x Male Club
* WP x Female Varsity
* WP x Male Varsity
* WP x Female Club
* WP x Male Club

Study Design and Procedures: The study will follow a randomized controlled parallel design over a two-year period. At the beginning of their training season, varsity (year one) and club athletes (year two) will be invited to participate in this 24-week study, consisting of an 8-week control condition (September to November) and a 16-week intervention condition (November to March).

Control Condition: During the 8-week control condition, participants will be instructed to follow their typical, habitual diet and training protocols. Seven-day food records will be completed by participants and assessed by a registered dietitian (RD) using the Keenoa online food tracker application in order to determine baseline dairy, calcium, and protein, intake levels in their habitual diets during the competitive season.

Intervention Condition: During the 16-week intervention condition, participants will be randomly assigned to either the GY or WP group. To monitor adherence, all participants will be asked to log their daily GY or WP intake.

Participants in the GY group will be instructed by the RD to consume 2 servings/day of 175 g commercially available GY (0% MF, flavoured, 130 calories, 17 g protein, 225 g calcium; e.g., OIKOS High Protein GY) for a total of 16 weeks. This serving amount has been used in the investigators' previous study in adolescent female soccer players, but slightly lower than in recreationally active adult males. For their convenience, the athletes will be provided with appropriate scoops to measure out 175 g of GY per serving of the larger 650 g commercially available, pre-packaged containers. Although it is recommended to consume the two servings morning and night, to increase ecological validity and strengthen the feasibility of the intervention, the timing of the servings will be flexible to facilitate the training and competition routines. For the same reasons, the athletes will be able to choose the flavour of their GY.

Participants in the WP group will follow a similar consumption schedule but will be instructed by the RD to consume two servings/day of 2/3 of a scoop of commercially available WP powder (flavoured, ~29 g, 120 calories, 19 g protein, 112.5 g calcium; e.g., PURE Whey Protein, Walmart) for a total of 16 weeks. The WP scoop will be dissolved in water (e.g., 1 g of WP isolate to 10 mL of water, as recommended by the manufacturer). This protein dose is similar to the previous dose in young swimmers and comparable to other studies in adults. Athletes will be provided with appropriately marked scoops (corresponding to 2/3 of the manufacturer scoop) to measure their single servings.

For the duration of both the GY and WP intervention condition (16 weeks), participants will be asked to maintain their habitual intakes (as per what they were doing in the control condition). That is, they will not be asked to stop any other protein supplementation they may have been taking during the control condition. The GY/WP servings during the intervention condition will be added to their habitual diet. Participants will be asked to track their daily dietary intake several times during the study (weeks 0, 8, 16, and 24), including all food, liquids, and supplements, using the Keenoa online food tracker application. Despite the added energy intake from the GY/WP, we do not expect any (significant) weight gain with the added ~300 calories per day due to the athletes' high energy expenditures.

Blood Samples: All participants will be instructed not to consume any food or liquids (except water, as needed) 8 hours prior to the time of their blood draw, not to exercise for 12 hours prior to the blood draw, and not to make any changes to their normal routines. A total of 10 mL of blood will be collected from an antecubital vein by a certified phlebotomist or registered nurse using a standard venipuncture technique at four timepoints: weeks 0, 8,16, and 24. All blood samples will be centrifuged at 1,405 x g at 4°C for 10 min. Serum and plasma will be aliquoted into pre-labeled Eppendorf tubes and stored at -80°C until analysis. The serum concentrations of markers and regulators of bone remodelling (osteocalcin, P1NP, CTX, OPG, sclerostin, RANKL, PTH), and the plasma concentrations of inflammatory cytokines (IL6, IL10, TNFα), sex hormones (estrogen, testosterone) and growth factors (IGF-1) will be measured in duplicate using commercially available ELISA kits.

Bone Properties: Transaxial quantitative ultrasound (QUS; Sunlight Omnisense™ 7000S, Sunlight Medical, Israel) will be used at weeks 0, 8, 16, and 24 to assess bone strength by measuring the speed of sound (SOS; m/s) along the bone at the distal 1/3 of the radius and at the mid-tibia of the dominant limbs, as previously described. The strength of bone is determined by the shortest time elapsed between the transmission and reception of the signal transmitted, with faster transmissions reflecting stronger bone. QUS can be used for the assessment of bone strength and is particularly suited for studies in healthy populations as it is portable, relatively inexpensive, and non-invasive (no radiation exposure). Because QUS measures the SOS along the bone it is not affected by bone size, thus allowing for comparisons between participants of different sizes. QUS has been previously used by the principal investigator and others to demonstrate the effect of exercise training or physical activity on various bones and in different age groups, including children.

Body Composition: Body mass (kg) and body composition will be measured using bioelectrical impedance analysis (BIA; InBody520 bioelectrical impedance analysis system following standard procedures.

Dietary Assessment: Participants' dietary intake, including energy intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded at weeks 0, 8, 16, and 24 using the Keenoa food application. Using the same application, participants will be asked to log their daily GY or WP intake in order to monitor adherence. In addition, participants' knowledge of nutrition will be assessed at the beginning (week 0) and completion of the study (week 24) using the self-reported 97-item GeSNK. The GeSNK encompasses 64 items assessing general and sport-specific nutrition knowledge, with the aim of exploring knowledge regarding macro- and micronutrients in various food choices, and awareness of diet-health associations, knowledge of fluid replacement, supplement intake, and food choices in regard to sport recovery meals. The GeSNK will be completed online along with the medical screening questions used to screen for inclusion criteria.

Training Volume and Physical Activity: Training logs will be collected from participants and coaches every week throughout the study. In addition, leisure-time physical activity will be assessed using the GSLTPAQ modified for the purpose of this study. The GSLTPAQ evaluates leisure-time physical activity using indicators of the intensity of exertion as light, moderate, vigorous, or very vigorous. Weekly physical activity metabolic equivalents are estimated based on the number of 15 min blocks at each intensity level multiplied by assumed energy consumption values. The GSLTPAQ is a standardized tool that has been demonstrated to be valid and reliable in children, adolescents, and adults.

Statistical Analysis: The data analysis with all ages combined using age and/or training volume as covariates will be performed leading to at least one additional publication and presentation. Prior to analysis, all variables will be tested for normality by visual inspection of histograms and z-scores (± 3) and by assessing the skewness and kurtosis (± 3). For dependent variables that are normally distributed, a series of two-way repeated measures analysis of variances with sex or age/training volume as covariates (RM-ANCOVAs) will be used to examine changes over time with main effects and interactions for the intervention conditions (GY vs WP) and time (0, 8, 16, and 24 weeks) on body composition and biochemical markers. In the event of a significant interaction or a main effect for time, posthoc pairwise comparisons will be performed with Bonferroni adjustment for multiple comparisons. If the assumption of sphericity is violated, the Greenhouse Geisser correction factor will be used. Dependent variables that may not be normally distributed will be log-transformed before the analysis. The significance level will be set at p <0.05.

Sample Size: Using G*Power analysis for an RM-ANCOVA (2 intervention groups, 4 timepoints, sex as covariate), we calculated that a total sample size of n = 36 (i.e., 18 per intervention group) would be required to detect a medium effect of partial η2 = 0.06 with a power of (1-β) = 0.90, and a probability level of p = 0.05. Thus, the proposed total of 40 participants (40 varsity and 40 club athletes) is more than adequate to detect significant effects and interactions, while allowing for a 20% attrition rate.

ELIGIBILITY:
Inclusion Criteria:

* Competitive youth or varsity athletes

Exclusion Criteria:

* Presence of injury
* Inability to participate in practices
* Allergy to dairy foods/dairy protein or
* Diagnosis with lactose intolerance

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Osteocalcin | Baseline (week 0)
  Morning, fasted, resting serum levels of the bone remodelling marker osteocalcin (ng/ml)
Osteocalcin | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of the bone remodelling marker osteocalcin (ng/ml)
Osteocalcin | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of the bone remodelling marker osteocalcin (ng/ml)
Osteocalcin | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of the bone remodelling marker osteocalcin (ng/ml)
Amino-terminal propeptide of type I collagen (P1NP) | Baseline (week 0)
  Morning, fasted, resting serum levels of bone formation marker P1NP (pg/ml)
Amino-terminal propeptide of type I collagen (P1NP) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone formation marker P1NP (pg/ml)
Amino-terminal propeptide of type I collagen (P1NP) | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone formation marker P1NP (pg/ml)
Amino-terminal propeptide of type I collagen (P1NP) | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone formation marker P1NP (pg/ml)
Osteoprotegerin (OPG) | Baseline (week 0)
  Morning, fasted, resting serum levels of bone formation regulator OPG (pg/ml)
Osteoprotegerin (OPG) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone formation regulator OPG (pg/ml)
Osteoprotegerin (OPG) | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone formation regulator OPG (pg/ml)
Osteoprotegerin (OPG) | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone formation regulator OPG (pg/ml)
C-telopeptides of type I collagen (CTX) | Baseline (week 0)
  Morning, fasted, resting serum levels of bone resorption marker CTX (ng/ml)
C-telopeptides of type I collagen (CTX) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone resorption marker CTX (ng/ml)
C-telopeptides of type I collagen (CTX) | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone resorption marker CTX (ng/ml)
C-telopeptides of type I collagen (CTX) | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone resorption marker CTX (ng/ml)
Sclerostin | Baseline (week 0)
  Morning, fasted, resting serum levels of bone resorption regulator sclerostin (pg/ml)
Sclerostin | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone resorption regulator sclerostin (pg/ml)
Sclerostin | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone resorption regulator sclerostin (pg/ml)
Sclerostin | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone resorption regulator sclerostin (pg/ml)
Receptor activator of nuclear factor kappa-Β ligand (RANKL) | Baseline (week 0)
  Morning, fasted, resting serum levels of bone resorption regulator RANKL (pg/ml)
Receptor activator of nuclear factor kappa-Β ligand (RANKL) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone resorption regulator RANKL (pg/ml)
Receptor activator of nuclear factor kappa-Β ligand (RANKL) | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone resorption regulator RANKL (pg/ml)
Receptor activator of nuclear factor kappa-Β ligand (RANKL) | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone resorption regulator RANKL (pg/ml)
Parathyroid hormone (PTH) | Baseline (week 0)
  Morning, fasted, resting serum levels of bone related hormone PTH (pmol/L)
Parathyroid hormone (PTH) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting serum levels of bone related hormone PTH (pmol/L)
Parathyroid hormone (PTH) | Middle of intervention period (week 16)
  Morning, fasted, resting serum levels of bone related hormone PTH (pmol/L)
Parathyroid hormone (PTH) | Completion of intervention period (week 24)
  Morning, fasted, resting serum levels of bone related hormone PTH (pmol/L)
Interleukin-6 (IL6) | Baseline (week 0)
  Morning, fasted, resting plasma levels of the inflammatory cytokine IL6 (pg/ml)
Interleukin-6 (IL6) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of the inflammatory cytokine IL6 (pg/ml)
Interleukin-6 (IL6) | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of the inflammatory cytokine IL6 (pg/ml)
Interleukin-6 (IL6) | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of the inflammatory cytokine IL6 (pg/ml)
Interleukin-10 (IL10) | Baseline (week 0)
  Morning, fasted, resting plasma levels of the anti-inflammatory cytokine IL10 (pg/ml)
Interleukin-10 (IL10) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of the anti-inflammatory cytokine IL10 (pg/ml)
Interleukin-10 (IL10) | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of the anti-inflammatory cytokine IL10 (pg/ml)
Interleukin-10 (IL10) | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of the anti-inflammatory cytokine IL10 (pg/ml)
Tumour necrosis factor-alpha (TNFα) | Baseline (week 0)
  Morning, fasted, resting plasma levels of the pro-inflammatory cytokine TNFα (pg/ml)
Tumour necrosis factor-alpha (TNFα) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of the pro-inflammatory cytokine TNFα (pg/ml)
Tumour necrosis factor-alpha (TNFα) | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of the pro-inflammatory cytokine TNFα (pg/ml)
Tumour necrosis factor-alpha (TNFα) | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of the pro-inflammatory cytokine TNFα (pg/ml)

SECONDARY OUTCOMES:
Insulin-like growth factor 1 (IGF1) | Baseline (week 0)
  Morning, fasted, resting plasma levels of IGF1 (ng/ml)
Insulin-like growth factor 1 (IGF1) | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of IGF1 (ng/ml)
Insulin-like growth factor 1 (IGF1) | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of IGF1 (ng/ml)
Insulin-like growth factor 1 (IGF1) | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of IGF1 (ng/ml)
Testosterone | Baseline (week 0)
  Morning, fasted, resting plasma levels of testosterone (pg/ml) will be measured in male athletes
Testosterone | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of testosterone (pg/ml) will be measured in male athletes
Testosterone | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of testosterone (pg/ml) will be measured in male athletes
Testosterone | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of testosterone (pg/ml) will be measured in male athletes
Estrogen | Baseline (week 0)
  Morning, fasted, resting plasma levels of estrogen (pg/ml) will be measured in female athletes
Estrogen | End of control period and pre-intervention (week 8)
  Morning, fasted, resting plasma levels of estrogen (pg/ml) will be measured in female athletes
Estrogen | Middle of intervention period (week 16)
  Morning, fasted, resting plasma levels of estrogen (pg/ml) will be measured in female athletes
Estrogen | Completion of intervention period (week 24)
  Morning, fasted, resting plasma levels of estrogen (pg/ml) will be measured in female athletes
Body mass | Baseline (week 0)
  Body mass (kg) will be measured using Bioelectrical Impedance
Body mass | End of control period and pre-intervention (week 8)
  Body mass (kg) will be measured using Bioelectrical Impedance
Body mass | Middle of intervention period (week 16)
  Body mass (kg) will be measured using Bioelectrical Impedance
Body mass | Completion of intervention period (week 24)
  Body mass (kg) will be measured using Bioelectrical Impedance
Fat mass | Baseline (week 0)
  Fat mass (kg) will be measured using Bioelectrical Impedance
Fat mass | End of control period and pre-intervention (week 8)
  Fat mass (kg) will be measured using Bioelectrical Impedance
Fat mass | Middle of intervention period (week 16)
  Fat mass (kg) will be measured using Bioelectrical Impedance
Fat mass | Completion of intervention period (week 24)
  Fat mass (kg) will be measured using Bioelectrical Impedance
Lean mass | Baseline (week 0)
  Lean mass (kg) will be measured using Bioelectrical Impedance
Lean mass | End of control period and pre-intervention (week 8)
  Lean mass (kg) will be measured using Bioelectrical Impedance
Lean mass | Middle of intervention period (week 16)
  Lean mass (kg) will be measured using Bioelectrical Impedance
Lean mass | Completion of intervention period (week 24)
  Lean mass (kg) will be measured using Bioelectrical Impedance
Body fat percentage | Baseline (week 0)
  Body fat percentage (%) will be measured using Bioelectrical Impedance Analysis
Body fat percentage | End of control period and pre-intervention (week 8)
  Body fat percentage (%) will be measured using Bioelectrical Impedance Analysis
Body fat percentage | Middle of intervention period (week 16)
  Body fat percentage (%) will be measured using Bioelectrical Impedance Analysis
Body fat percentage | Completion of intervention period (week 24)
  Body fat percentage (%) will be measured using Bioelectrical Impedance Analysis
Height | Baseline (week 0)
  Height (cm) will be measured using a stadiometer
Height | End of control period and pre-intervention (week 8)
  Height (cm) will be measured using a stadiometer
Height | Middle of intervention period (week 16)
  Height (cm) will be measured using a stadiometer
Height | Completion of intervention period (week 24)
  Height (cm) will be measured using a stadiometer
Bone Properties | Baseline (week 0)
  Bone speed of sound (m/s) will be measured with transaxial quantitative ultrasound
Bone Properties | End of control period and pre-intervention (week 8)
  Bone speed of sound (m/s) will be measured with transaxial quantitative ultrasound
Bone Properties | Middle of intervention period (week 16)
  Bone speed of sound (m/s) will be measured with transaxial quantitative ultrasound
Bone Properties | Completion of intervention period (week 24)
  Bone speed of sound (m/s) will be measured with transaxial quantitative ultrasound
Dietary intake (kcal/day) | Baseline (week 0)
  Participants' dietary intake, including energy intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded using the Keenoa food application. Using the same application, participants will be asked to log their GY or WP intake in order to monitor adherence.
Dietary intake (kcal/day) | End of control period and pre-intervention (week 8)
  Participants' dietary intake, including energy intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded using the Keenoa food application. Using the same application, participants will be asked to log their GY or WP intake in order to monitor adherence.
Dietary intake (kcal/day) | Middle of intervention period (week 16)
  Participants' dietary intake, including energy intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded using the Keenoa food application. Using the same application, participants will be asked to log their GY or WP intake in order to monitor adherence.
Dietary intake (kcal/day) | Completion of intervention period (week 24)
  Participants' dietary intake, including energy intake, as well as macronutrient, micronutrient, vitamin, and supplement intakes will be recorded using the Keenoa food application. Using the same application, participants will be asked to log their GY or WP intake in order to monitor adherence.
Energy expenditure (kcal/week) | Baseline (week 0)
  Leisure-time physical activity will be assessed using the GSLTPAQ modified for the purpose of this study
Energy expenditure (kcal/week) | End of control period and pre-intervention (week 8)
  Leisure-time physical activity will be assessed using the GSLTPAQ modified for the purpose of this study
Energy expenditure (kcal/week) | Middle of intervention period (week 16)
  Leisure-time physical activity will be assessed using the GSLTPAQ modified for the purpose of this study
Energy expenditure (kcal/week) | Completion of intervention period (week 24)
  Leisure-time physical activity will be assessed using the GSLTPAQ modified for the purpose of this study
Training volume (hours/week) | Baseline (week 0)
  Training logs will be collected from participants and coaches
Training volume (hours/week) | End of control period and pre-intervention (week 8)
  Training logs will be collected from participants and coaches
Training volume (hours/week) | Middle of intervention period (week 16)
  Training logs will be collected from participants and coaches
Training volume (hours/week) | Completion of intervention period (week 24)
  Training logs will be collected from participants and coaches
Nutrition knowledge | Baseline (week 0)
  Participants' knowledge of nutrition will be assessed using the self-reported 97-item General and Sport-Specific Nutrition Knowledge Questionnaire (GeSNK)
Nutrition knowledge | Completion of intervention period (week 24)
  Participants' knowledge of nutrition will be assessed using the self-reported 97-item General and Sport-Specific Nutrition Knowledge Questionnaire (GeSNK)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Klentrou, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada